CLINICAL TRIAL: NCT02228746
Title: Effect of the Alpha-galacto-oligasaccharides on Weight Loss in Overweight or Moderately Obeses Adults : A Randomized Controlled Double Blinded Trial Versus Placebo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olygose (Industry)
Collaborators: Institute of Cardiometabolism and Nutrition, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-A01610--43
Record Dates: First submitted 2014-04-28; First posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Randomized Versus Placebo; Controlled; Double Blind

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alpha-galacto-oliosaccharides (Experimental)
  Interventions: Dietary Supplement: Alpha-galacto-oligosaccharides
- Placebo (Placebo Comparator)

INTERVENTIONS:
Dietary Supplement: Alpha-galacto-oligosaccharides — 6g of alpha-galacto-oligosaccharides in a 100 mL flavored drink
  Arms: Alpha-galacto-oliosaccharides

SUMMARY:
Clinical intervention on overweight or moderately obeses adults. The objective of this trial is to demonstrate the superior eficacy of Alphagos to placebo on weight loss during a low-calorie diet of 12 weeks. The superiority is judged on body weight. Change in cardiometabolic risk factors through the intervention have been evaluated as secondary endpoints

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index > or equal 25 and < 35
* Use of effective contraception in women of childbearing age

Exclusion Criteria:

* Pregnant women (positive pregnancy test) or breastfeeding
* Anti-hypertensive or cholesterol treatment
* HIV infection or HCV
* Hepatic and/or severe renal failure
* Heart attack within 6 months prior the selection
* Heart failure known
* Inflammatory disease known
* Cancer or have had cancer within 3 years prior to the study except for basal cell skin cancers
* Diabetes defined by blood glucose greater than or equal to 1.26 g/L
* Gastrointestinal disease known
* Bariatric surgery

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Body weight (kg) between day 0 and week 12 | Day 0, Day 7, Month 1, Month 2, Month 3

SECONDARY OUTCOMES:
Feeding behaviour | Between day 0 and week 12
  Changes in feeding behaviour will be studied by :
  * visual analogue scales rating for hunger, satiety, fullness, desire to eat, prospective consumption during preload-test meal paradigm (standardized breakfast and lunch test)
  * level of circulating peptides involved in the regulation of controlling food intake during a kinetic after a standardized breakfast (samples 30, 60, 120, 180 and 240 min after the start of standardized breakfast)
  * food intake during the lunch test
Lean body mass | Between day 0 and week 12
Waist circumference | Day 0, day 7, Month1, Month 2, Month 3
Hip circumference | Day 0, Day 7, Month 1, Month 2, Month 3
Waist to hip circumference ratio | Between Day 0 and week 12
Body Fat | Day 7, Month 3

OTHER OUTCOMES:
Body Mass Index (BMI) | between Day 0 and week 12
arterial systolic and diastolic pressures | between day 0 and week 12
Morphological, inflammatory and metabolic characteristics of adipose tissue sampled from the abdominal region | between day 0 and week 12
  Adipocyte size and diameter, secretion profile of subcutaneous adipose tissue, gene expression profile of adipose tissue, lipolytic response and energy metabolism
Components of the intestinal commensal microbiota | between day 0 and week 12
Lipid Profile | Day 0, Week 12
Markers of systemic inflammation | Day 0, Week 12
Glycemic profile | Day 0, Week 12
Circulating adipokines | Day 0, Week 12
Hemostatic factors associated with cardiovascular risks | Day 0, Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Investigation Clinique Paris-Est/ Bâtiment Antonin Gosset Hôpital de la Pitié Salpêtrière- 56 Boulevard Vincent Auriol, Paris, France